CLINICAL TRIAL: NCT04848922
Title: The Effect of Hot Showers on Postpartum Fatigue, Mood and Comfort In Women Giving Vaginal Birth: A Randomized Controlled Trial
Brief Title: Hot Showers on Postpartum Fatigue, Mood and Comfort In Women Giving Vaginal Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Rabia Atilla, Lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OHU_Ratilla; TDK-2018-8319 (Other Grant/Funding Number: Erciyes University); 2017/532 (Other: Erciyes University)
Record Dates: First submitted 2021-04-10; First posted 2021-04-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Fatigue; Comfort; Mood; Postpartum Care
Keywords: Postpartum Maternal Health; Hot Shower; Fatigue; Comfort; Mood; Nursing-Midwifery Care
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Took a hot shower intervention and usual care.
  Interventions: Other: Hot shower intervention
- Control Group (No Intervention): No intervention other than usual care.

INTERVENTIONS:
Other: Hot shower intervention — Intervention group took a shower in a standing position at a water temperature of 37-41°C for 10-20 minutes between 6 and 12 hours after vaginally birth.
  Arms: Intervention Group

SUMMARY:
The aim of this study to determine the effect of hot showers on postpartum fatigue, mood and comfort in women giving vaginal birth. 136 women, who were between 6 and 12 hours postpartum, were assigned to intervention and control groups by computer randomization. Visual Similarity Scale for Fatigue, Visual Analogue Scale, Postpartum Comfort Questionnaire and Brief Mood Insight Scale were used to collect data. The women in the intervention group were allowed to take a shower in a standing position at a water temperature of 37-41°C for 10-20 minutes. In the control group, routine care was provided.

DETAILED DESCRIPTION:
Evidence has been limited on the effect of hot showers on postpartum fatigue, mood, and comfort in women giving vaginal birth. This study aimed to determine such effects in a randomized controlled trial conducted in a hospital in Turkey. Participants were recruited from a hospital located in the Nigde province in the Central Anatolia region in Turkey. The data of the research were collected between 9 April 2018 and 13 February 2019.

Puerperal women who had given birth in vaginal way and who were in the maternity ward of the hospital and who were between 6 and 12 hours postpartum were included in the study. The computer-generated randomization list was prepared by an independent biostatistician using the PASS program (PASS 11.0.4, NCSS, LL. Kaysville, Utah, and USA). Women who met the inclusion criteria were randomized into intervention group (IG) and the control group (CG) based on age and parity status (through one-to-one matching) by computer. A total of 128 volunteers, 64 in each group, were included in the study in order to be able to determine an effect size of 0.5 between the two groups, with an error risk of α = 0.05 and 80% power ratio to represent the medium effect size using Cohen's (1988) effect size. However, it was predicted that there might be withdrawals during the study, and 136 women, 68 in each group, were included in the study.

Puerperium Introduction Form (PIF), Puerperium Follow-Up Form (PFF), Visual Similarity Scale for Fatigue (VSSF), Visual Analogue Scale for Fatigue and Disomfort (VAS-F and VAS-D), Postpartum Comfort Questionnaire (PPCQ) and Brief Mood Insight Scale (BMIS) were used to collect data.

At the first interview, 6 and 12 hours postpartum, PIF, VAS for fatigue and discomfort, and VSSF were filled in for the puerperal women in the Intervention Group (IG) and Control Group (CG). In the CG, women were provided routine care practices in the postnatal care unit of the hospital. In the IG, in addition to the routine care practices of the clinic, a hot shower at a standing position was provided. The temperature of the water was adjusted according to the preferences of the women to between 37 and 41 °C with a digital shower thermometer, and the women were allowed to shower for 10-20 minutes in a standing position. After the shower procedures, the information on and individual views of the puerperal women were recorded in the PFF. One hour after the completion of the hot shower procedure, the VAS for fatigue and discomfort, the VSSF, the PPCQ, and BMIS were filled in for the final test.

Data analyses were conducted using IBM SPSS 25.0 software. Chi-square and t statistical tests were used to to determine whether the socio-demographic and obstetric characteristics. For numerical variable comparisons between groups were evaluated using two independent samples t-test for variables that provide normal distribution assumption, and the Mann-Whitney U test for variables that do not provide a normal distribution assumption. For numerical variables, the comparisons of the groups over time were made with Repeated Measures ANOVA. The Bonferroni test was used as a multiple comparison test. In cases where p <.05, the difference between groups was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Puerperal women who were aged 19 and over,
* Educated to at least primary school level,
* Have a vaginal delivery,
* To be between 6 and 12 hours postpartum duration ,
* Having a single and healthy newborn,
* Mobilized.

Exclusion Criteria:

* Puerperal women with a history of chronic illness
* Puerperal women with a history of psychiatric illness
* Any risk diagnosed pregnancy (such as oligohydramnios, preeclampsia, heart disease, diabetes, placenta previa)
* Any complications related to the mother and baby in birth period (dystocia,operative birth, bleeding, hypertension),
* Any complications related to the mother and baby in the postpartum period (bleeding, hypo-hypertension, babies taken to the neonatal intensive care unit, a body temperature of 38 °C or above, positive Homan's sign etc.).
* Have a body mass index of 40 or above
* Have Anemic

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Fatigue Scores | At baseline and an hour after intervention, fatigue was assessed.
  Fatigue assessed using by The Visual Similarity Scale for Fatigue (VSSF) and Visual Analog Scale (VAS-F).
  The Visual Similarity Scale for Fatigue (VSSF) consists of 18 items in two sub-dimensions, comprising fatigue (13 items) and energy (5 items) sub-dimensions. The scale consists of 10-cm horizontal lines that contain positive expressions at one end and negative expressions at the other end. The intersection point at the marked location is evaluated objectively by measuring it with a ruler separately for each question. The score range in the sub-dimension of fatigue is 0-130.
  Visual Analog Scale (VAS-F) is a scale on a 10 cm long vertical line with two ends named differently (0 = I am not tired and 10 = I am extremely tired). The distance between the marked point and the lowest end of the line (0 = I'm not tired) is measured in centimeters and the numerical value found indicates the patient's fatigue severity.
Comfort Scores | PPCQ was assessed an hour after intervention.
  Comfort assessed using by Postpartum Comfort Questionnaire (PPCQ). Postpartum Comfort Questionnaire (PPCQ) which is a five-point likert type scale, has 34 items and the total score is 34-170. The scale has three sub-dimensions: "physical, psycho-spiritual and sociocultural". The comfort score is expressed as the average value, obtained by dividing the total score by the number of items. The average value found is shown in a distribution of 1 (low comfort) to 5 (high comfort).
Discomfort Scores | VAS-D was assessed at baseline and an hour after intervention.
  Discomfort assessed using by Visual Analog Scale for Discomfort (VAS-D). Visual Analog Scale for Discomfort (VAS-D) is a scale on a 10 cm long vertical line with two ends named differently (0 = No discomfort and 10 = Extremely discomfort). The distance between the marked point and the lowest end of the line (0 = No discomfort) is measured in centimeters and the numerical value found indicates the patient's discomfort severity.
Mood Scores | BMIS was assessed an hour after intervention.
  Brief Mood Insight Scale (BMIS) which is likert type scale, has 16 items with four scores (1 (absolutely not) -4 (absolutely feel)) and the total score is 8-32. High scores for both subscales indicate high positive or negative mood.

SECONDARY OUTCOMES:
Energy Scores | At baseline and an hour after intervention, energy was assessed.
  The Visual Similarity Scale for Fatigue (VSSF) consists of 18 items in two sub-dimensions, comprising fatigue (13 items) and energy (5 items) sub-dimensions. The scale consists of 10-cm horizontal lines that contain positive expressions at one end and negative expressions at the other end. The intersection point at the marked location is evaluated objectively by measuring it with a ruler separately for each question. The score range 0-50 in the sub-dimension of energy.

OTHER OUTCOMES:
Opinions about Postpartum Hot Showers İntervention | PFF was assessed an hour after intervention
  Puerperium Follow-Up Form (PFF): This is a form consisting of a total of three questions, in which are recorded the individual views of members of the intervention group regarding the duration of the shower procedure and the negative effects that may have been experienced. In addition, there is a question regarding the control group's views on postpartum shower application.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No